CLINICAL TRIAL: NCT04008069
Title: A Phase II, Single-Site, Double-Blind, Placebo-Controlled Randomized Withdrawal Study Assessing the Efficacy and Safety of Sarilumab in Patients With Glucocorticoid-Dependent Sarcoidosis
Brief Title: Sarilumab in Patients With Glucocorticoid-Dependent Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew C. Baker, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 48375
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Sarcoidosis
Keywords: glucocorticoid-dependent
MeSH Terms: conditions — Sarcoidosis | interventions — sarilumab

STUDY DESIGN:
Intervention Model Description: All subjects will all receive sarilumab 200 mg subcutaneously every two weeks for the first 16 weeks of the study. At Week 16, those patients who were able to successfully taper off of prednisone will then be assigned randomly to receive either sarilumab 200 mg subcutaneously every two weeks (study drug) or placebo subcutaneously for an additional 12 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study doctor and personnel will not know whether you are assigned to the sarilumab group or the placebo group after Week 16.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open-Label Sarilumab (pre-randomization) (Experimental): On entering the study, all participants receive open-label sarilumab every two weeks for 16 weeks.
  Interventions: Drug: Sarilumab
- Double-Blind Sarilumab (post-randomization) (Experimental): After completing the open-label period, participants are randomized in blinded fashion to receive sarilumab every two weeks for 12 weeks.
  Interventions: Drug: Sarilumab
- Double-Blind Placebo (post-randomization) (Placebo Comparator): After completing the open-label period, participants are randomized in blinded fashion to receive placebo every two weeks for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarilumab — Sarilumab 200 mg administered subcutaneously
  Other Names: Kevzara
  Arms: Double-Blind Sarilumab (post-randomization); Open-Label Sarilumab (pre-randomization)
Drug: Placebo — Placebo administered subcutaneously
  Arms: Double-Blind Placebo (post-randomization)

SUMMARY:
The purpose of this study is to compare the effectiveness and the safety of sarilumab in patients with glucocorticoid-dependent sarcoidosis.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectivness and the safety of sarilumab in patients with glucocorticoid-dependent sarcoidosis. To demonstrate that sarilumab treatment will be effective for inducing and maintaining glucocorticoid-free remission in male or female patients with biopsy proven active, glucocorticoid-dependent sarcoidosis affecting the lungs, lymph nodes, liver, kidneys, spleen, bone, soft tissues, skin, and/or eyes.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven non-caseating granulomas consistent with sarcoidosis
* negative infectious studies including AFB and fungal stains, and with compatible clinical and/or radiographic manifestations of sarcoidosis.
* Involvement of the lungs (stage II or III pulmonary sarcoidosis), lymph nodes, liver, kidneys, spleen, bone, soft tissues, skin, and/or eyes.
* At least one active manifestation, defined by the need for ongoing glucocorticoid treatment to control a sign or symptom of sarcoidosis, which requires treatment with prednisone (or equivalent corticosteroid) ≥ 10 mg and ≤ 60 mg daily (i.e. glucocorticoid dependence), with stable dosing for ≥ 28 days prior to baseline.
* patients taking a glucocorticoid other than prednisone, will be changed to prednisone at the equivalent dose and take this daily for ≥ 14 days prior to baseline.
* DMARDs including methotrexate, leflunomide, azathioprine, mycophenolate mofetil, and/or anti-malarials (i.e. hydroxychloroquine) permitted must be stable for ≥ 28 days prior to baseline and remain stable during follow-up.

Exclusion Criteria:

* Stage IV pulmonary sarcoidosis.
* Central nervous system sarcoidosis.
* Cardiac sarcoidosis.
* Prior treatment with an anti-IL-6 therapy.
* Treatment with a biologic agent including rituximab, belimumab, TNF inhibitors, abatacept, or IL-17 inhibitors administered within 28 days prior to baseline (6 months for rituximab).
* Treatment with cyclophosphamide within 3 months prior to baseline.
* Treatment with prednisone < 10 mg or > 60 mg daily.
* Known hypersensitivity or allergy to the study drug.
* History of, or current, inflammatory or autoimmune disease other than sarcoidosis which would present a safety issue or confound interpretation of the data.
* Prior or current history of other significant concomitant illness that, according to the investigator's judgment, would adversely affect the patient's participation in the study. These include, but are not limited to, cardiovascular (including stage III or IV cardiac failure according to the New York Heart Association classification), neurological (including demyelinating disease), active infectious diseases, or history of diverticulitis or gastrointestinal perforation.
* Patients currently pregnant or breast-feeding.
* Women of childbearing potential (WOCBP) who are unwilling to utilize adequate contraception and unwilling to not become pregnant during the full course of the study (must be willing to be tested for pregnancy). Adequate contraceptive measures include oral contraceptives (continuous use, as per prescription, for 2 or more cycles prior to screening), intrauterine devices, contraceptive sponges, condoms or diaphragms plus foam, or jelly, or surgical procedures such as bilateral tubal ligation or vasectomy in partner.
* Administration of a live/attenuated vaccine within 30 days.
* Evidence of active tuberculosis, HIV, or hepatitis B or C infection.
* History of cancer other than non-melanoma skin cancer.
* Patients with any of the following laboratory abnormalities at the screening visit: hemoglobin <8.5 g/dL, white blood cells <3000/mm3, neutrophils <2000/mm3, platelet count <150,000 cells/mm3, aspartate aminotransferase (AST) or ALT >1.5 x ULN, and/or bilirubin (total) above the upper limit of normal (unless Gilbert's disease has been determined by genetic testing and documented).
* Presence of severe uncontrolled hypercholesterolemia (>350 mg/dL, 9.1 mmol/L) or hypertriglyceridemia (>500 mg/dL, 5.6 mmol/L) at screening or baseline.
* Patients with calculated creatinine clearance <30 mL/minute (using Cockroft-Gault formula).
* History of alcohol or drug abuse within 5 years prior to the screening visit.
* Participation in any clinical research study evaluating another investigational drug or therapy within 5 half-lives or 60 days of first investigational medicinal product (IMP) administration, whichever is longer.
* Any patient who has had surgery within 4 weeks prior to the screening visit or with planned surgery during the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Baker, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Baker MC, Horomanski A, Wang Y, Liu Y, Parsafar S, Fairchild R, Mooney JJ, Raj R, Witteles R, Genovese MC. A double-blind, placebo-controlled, randomized withdrawal trial of sarilumab for the treatment of glucocorticoid-dependent sarcoidosis. Rheumatology (Oxford). 2024 May 2;63(5):1297-1304. doi: 10.1093/rheumatology/kead373. PMID 37471590

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixteen participants were screened, fifteen met eligibility criteria and were allocated to treatment.
Groups:
- Open-Label Sarilumab (Pre-randomization): On entering the study, all participants receive open-label sarilumab (200 mg administered subcutaneously) every two weeks for 16 weeks.
- Double-Blind Sarilumab (Post-randomization): After completing the open-label period, participants are randomized to receive sarilumab (200 mg administered subcutaneously) every two weeks for 12 weeks.
- Double-Blind Placebo (Post-randomization): After completing the open-label period, participants are randomized receive placebo every two weeks for 12 weeks.
Period: Open-Label Period
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Started | 15 | 0 | 0
Completed Treatment up to Week 16 | 10 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Period: Randomized-Withdrawal Period
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Started | 0 | 2 | 8
Completed Treatment With Study Drug | 0 | 1 | 5
Completed | 0 | 1 | 5
Not Completed | 0 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who enter the study, to receive open-label sarilumab every two weeks for 16 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.51)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 4
  ≥ 50 Years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Sarcoidosis Flare (Flare-Free Survival)
Description: The primary outcome was flare-free survival of sarilumab-treated patients compared to placebo-treated controls. Patients will be considered to have flared if they receive rescue medication including increased glucocorticoids, or if they discontinue the study treatment in order to start a different therapy.
Time Frame: Week 16 to Week 28
Population: Assessed in participants in the randomized-withdrawal period
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Sarilumab (Post-randomization): After completing the open-label period, participants are randomized to receive sarilumab every two weeks for 12 weeks.
Arm/Group | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 2 | 8
Participants | 2 | 7

2. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted
Description: FVC is a pulmonary function test, and is defined as the volume of air that can forcibly be blown out after taking a full breath. FVC% predicted is defined as FVC% of the patient divided by the average FVC% in the population for any person of similar age, sex and body composition.
Time Frame: Baseline and week 16
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: FVC % predicted
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
FVC % predicted
  Baseline | 92.1 (19.8) | 113 (14.9) | 95.9 (17.3)
  Change at week 16: number analyzed (Participants) | 13 | 1 | 8
  Change at week 16 | -2.69 (4.89) | -11.0 (NA) — Not calculable for n of 1 | -1.38 (4.78)

3. Secondary Outcome: Change From Baseline in Hemoglobin-corrected Diffusing Capacity for Carbon Monoxide (DLCO) Percent Predicted
Description: DLCO is a pulmonary function test, and measures the partial pressure difference between inspired and expired carbon monoxide. DLCO% predicted is defined as DLCO% of the patient divided by the average DLCO% in the population for any person of similar age, sex and body composition.
Time Frame: Baseline, and week 16
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: DLCO % predicted
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 1 | 8
DLCO % predicted
  Baseline | 92.6 (21.4) | 90 (NA) — Not calculable for n of 1 | 93.5 (22.8)
  Change at week 16: number analyzed (Participants) | 15 | 0 | 8
  Change at week 16 | -14.8 (23.5) |  | -18.4 (28.9)

4. Secondary Outcome: Change in Pulmonary Function (FEV1) Percent Predicted
Description: FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height.
Time Frame: Baseline and week 16
Population: Data were collected during the open-label portion of the study only
Measure: Mean (Standard Deviation); unit: FEV1 % predicted
Arm/Group | Open-Label Sarilumab (Pre-randomization)
Number analyzed (Participants) | 15
FEV1 % predicted
  Baseline | 89.0 (19.86)
  Week 16 | 86.0 (18.25)

5. Secondary Outcome: Change From Baseline in Extrapulmonary Physician Organ Severity Tool (ePOST) Scale Score
Description: Physician and patient assessments assessed using the extrapulmonary physician organ severity tool (ePOST).
  Score Description:
  0: Not affected
  1. Slight
  2. Mild
  3. Moderate
  4. Moderate to severe
  5. Severe
  6. Very Severe 17 organ domains were rated and summed to create a total score (range 0-102, higher scores correspond with more severity).
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
score on a scale
  Baseline | 2.53 (3.00) | 7.50 (4.95) | 2.38 (1.85)
  Change at week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at week 16 | -0.57 (0.85) | -1.00 (1.41) | -0.75 (0.89)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at week 28 | -1.00 (1.10) | -2.00 (NA) — Not calculable for n of 1 | -0.80 (1.10)

6. Secondary Outcome: Change From Baseline in Physician Disease Activity Visual Analogue Scale (VAS)
Description: Physician rates patient's disease on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale (mm)
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
units on a scale (mm)
  Baseline | 48.0 (13.2) | 38.5 (20.5) | 45.3 (13.9)
  Change at week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at week 16 | -22.8 (22.2) | -13.0 (5.66) | -35.6 (11.3)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 8
  Change at week 28 | -31.8 (13.5) | -21.0 (NA) — Not calculable for n of 1 | -34.0 (13.9)

7. Secondary Outcome: Change From Baseline in Patient Disease Activity Visual Analogue Scale (VAS)
Description: Patient rates their disease on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale (mm)
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
units on a scale (mm)
  Baseline | 33.1 (22.7) | 11.5 (9.19) | 27.4 (23.6)
  Change at week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at week 16 | -4.86 (17.8) | 0.50 (7.78) | -11.1 (19.9)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at week 28 | -3.00 (34.4) | -5.00 (NA) — Not calculable for n of 1 | -2.50 (39.8)

8. Secondary Outcome: Change From Baseline in FACIT-F Score (Fatigue Scale)
Description: FACIT-F score
  Total score range: 0-52, lower scores correspond with more fatigue.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
score on a scale
  Baseline | 38.1 (10.8) | 51.0 (0) | 37.9 (12.4)
  Change at Week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at Week 16 | 1.86 (9.58) | -1.50 (2.12) | 5.62 (9.64)
  Change at Week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at Week 28 | 5.00 (12.8) | 0 (NA) — Not calculable for n of 1 | 6.25 (14.5)

9. Secondary Outcome: Number of Tender and Swollen Joints Per 68/66 Joint Evaluation
Description: The 66/68 Joint Count evaluates 68 joints for tenderness and pain with movement and 66 joints for swelling (hip joints can be evaluated for tenderness only, not for swelling.
  Joint evaluation score:
  0: Absent
  1: Present 9: Not applicable
Time Frame: Baseline, week 16, and week 28
Population: Participants who presented with inflammatory arthritis and with available data at each respective time point are included in the analysis.
Measure: Number; unit: joints
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 2 | 0 | 1
joints
  Baseline - tender joints | 20 |  | 18
  Baseline - swollen joints | 20 |  | 18
  Week 16 - tender joints | 4 |  | 0
  Week 16 - swollen joints | 18 |  | 16
  Week 28 - tender joints: number analyzed (Participants) | 1 | 0 | 1
  Week 28 - tender joints | 0 |  | 0
  Week 28 - swollen joints: number analyzed (Participants) | 1 | 0 | 1
  Week 28 - swollen joints | 8 |  | 8

10. Secondary Outcome: Sarcoidosis Activity and Severity Index for Cutaneous Sarcoidosis
Description: Sarcoidosis Activity and Severity Index evaluates 7 parameters on a 0 to 4 scale, summed for an overall scale score of 0 to 28 (higher values indicate higher activity/severity).
Time Frame: Baseline, week 16, and week 28
Population: Participants who presented with cutaneous sarcoidosis and with available data at each respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 3 | 0 | 2
score on a scale
  Baseline | 12.7 (9.29) |  | 9.5 (10.61)
  Week 16 | 16.7 (15.50) |  | 9.0 (11.31)
  Week 28: number analyzed (Participants) | 0 | 0 | 2
  Week 28 |  |  | 9.0 (11.31)

11. Secondary Outcome: Change in Size of Sarcoidosis Lesions
Time Frame: Baseline, week 16, and week 28
Population: Data were not collected for this outcome
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Serum Angiotensin Converting Enzyme
Description: ACE is a serum marker that is increased in sarcoidosis. ACE is produced by epithelioid cells that are derived from recently-activated macrophages in granulomas; thus, ACE is an appropriate representative of whole-body granuloma.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
U/L
  Baseline | 35.4 (23.5) | 63.0 (7.07) | 32.6 (26.6)
  Change at week 16: number analyzed (Participants) | 13 | 2 | 8
  Change at week 16 | 18.1 (24.6) | 55.5 (51.6) | 8.12 (11.9)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at week 28 | 7.17 (20.4) | 14.0 (NA) — Not calculable for n of 1 | 5.80 (22.5)

13. Secondary Outcome: Change From Baseline in Serum C-Reactive Protein (CRP)
Description: CRP is a protein made by the liver. The level of CRP increases when there's inflammation in the body.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
mg/dL
  Baseline | 0.52 (0.49) | 0.90 (1.13) | 0.41 (0.42)
  Change at week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at week 16 | -0.20 (0.76) | -0.90 (1.13) | -0.22 (0.53)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at week 28 | -0.20 (0.55) | 0 (NA) — Not calculable for n of 1 | -0.24 (0.61)

14. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is the rate at which red blood cells in anticoagulated whole blood descend in a standardized tube over a period of one hour.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Mean (Standard Deviation); unit: cells per hour
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
cells per hour
  Baseline | 9.33 (5.65) | 9.50 (2.12) | 10.9 (7.38)
  Change at week 16: number analyzed (Participants) | 14 | 2 | 8
  Change at week 16 | -3.00 (6.51) | -7.00 (1.41) | -3.43 (6.68)
  Change at week 28: number analyzed (Participants) | 6 | 1 | 5
  Change at week 28 | -2.00 (6.96) | -6.00 (NA) — Not calculable for n of 1 | -1.20 (7.46)

15. Secondary Outcome: Change in Prednisone Dose
Time Frame: Baseline, week 16, and week 28
Population: Data were not collected for this outcome
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Outside Normal Range
Description: Normal range as calculated by the local laboratory.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
Participants
  Baseline | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 14 | 2 | 8
  Week 16 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 6 | 1 | 5
  Week 28 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Aspartate Aminotransferase (AST) Outside Normal Range
Description: Normal range as calculated by the local laboratory.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
Participants
  Baseline | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 14 | 2 | 8
  Week 16 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 6 | 1 | 5
  Week 28 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Serum Creatinine Outside Normal Range
Description: Normal range as calculated by the local laboratory.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
Participants
  Baseline | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 14 | 2 | 8
  Week 16 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 6 | 1 | 5
  Week 28 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Urine Protein Outside Normal Range
Description: Normal range as calculated by the local laboratory.
Time Frame: Baseline, week 16, and week 28
Population: Participants with available data at each respective time point are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
Number analyzed (Participants) | 15 | 2 | 8
Participants
  Baseline | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 14 | 2 | 8
  Week 16 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 1 | 1 | 5
  Week 28 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | Open-Label Sarilumab (Pre-randomization) | Double-Blind Sarilumab (Post-randomization) | Double-Blind Placebo (Post-randomization)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 9/15 | 1/2 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Sarilumab (Pre-randomization) (N=15) | Double-Blind Sarilumab (Post-randomization) (N=2) | Double-Blind Placebo (Post-randomization) (N=8)
COVID-19 (Infections and infestations) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Sarilumab (Pre-randomization) (N=15) | Double-Blind Sarilumab (Post-randomization) (N=2) | Double-Blind Placebo (Post-randomization) (N=8)
Transaminitis (Investigations) | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Prolonged neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Ulcers aphthous oral (Gastrointestinal disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral vision defective (Eye disorders) | 1 | 0 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cervical radiculopathy (Reproductive system and breast disorders) | 0 | 0 | 1
Kappa light chain analysis increased (Investigations) | 1 | 0 | 0
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Creatinine kinase increased (Investigations) | 0 | 0 | 1
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pain in (r) hip (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Alcohol rehabilitation (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04008069/Prot_SAP_000.pdf